CLINICAL TRIAL: NCT01608945
Title: Prospective Randomized Study of Glucocorticoids in the Impact of the Liver Function and the Prognosis After Hepatectomy of HCC
Status: Suspended | Type: Observational
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, jian zhai, hepatic department, Eastern Hepatobiliary Surgery Hospital
Other Study IDs: EHBH112
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Some Studies Shows That the Steroid Can Reduce the Injury of the I/R of the Liver
Keywords: steroid; liver function; prognosis
MeSH Terms: interventions — Hydrocortisone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- steroid,liver function I/R
  Interventions: Drug: Hydrocortisone sodium succinate

INTERVENTIONS:
Drug: Hydrocortisone sodium succinate — 100mg/day

SUMMARY:
The major drawback of hepatic pedicle clamping is ischaemia-reperfusion injury with impairment of liver function. Perioperative steroid administration has been advocated to reduce liver damage. The aim of this prospective, randomized study was to determine whether steroid administration can reduce liver injury and impact the prognosis

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* diametre of the mass>3cm.
* hcc

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-04

PRIMARY OUTCOMES:
liver function | six months